CLINICAL TRIAL: NCT03825328
Title: A Phase II , Open-label , Investigator-initiated Trail of Sequential GEMOX/NS Chemotherapy in Patients With Untreated Pancreatic Cancer
Brief Title: A Trial of NS/GEMOX Chemotherapy in Patients With Untreated Pancreatic Cancer ( HZ-NS/GEMOX-PC )
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yanqiao Zhang (Other)
Responsible Party: Sponsor-Investigator, Yanqiao Zhang, Director of the hospital, Harbin Medical University
Organization: Harbin Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HZ-NS/GEMOX-PC
Record Dates: First submitted 2019-01-30; First posted 2019-01-31 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Albumin-Bound Paclitaxel; S 1 (combination); Oxaliplatin; Gemcitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chemotherapy (Experimental): Albumin-binding paclitaxel+S1 / gecitabine+oxaliplatin Interchanged every 2 cycles
  Interventions: Drug: Albumin-bound paclitaxel; Drug: S-1; Drug: Oxaliplatin; Drug: Gemcitabine

INTERVENTIONS:
Drug: Albumin-bound paclitaxel — Albumin-bound paclitaxel is paclitaxel formulated as albumin-bound nanoparticles with a mean particle size of approximately 130 nanometers.
Drug: S-1 — a combination preparation of tegafur, gimeracil, and oteracil potassium
Drug: Oxaliplatin — The compound features a square planar platinum(II) center. In contrast to cisplatin and carboplatin, oxaliplatin features the bidentate ligand 1,2-diaminocyclohexane in place of the two monodentate ammine ligands. It also features a bidentate oxalate group.
Drug: Gemcitabine — Gemcitabine is a synthetic pyrimidine nucleoside prodrug-a nucleoside analog in which the hydrogen atoms on the 2' carbon of deoxycytidine are replaced by fluorine atoms.

SUMMARY:
This is a Phase II , Open-label , Investigator-initiated Trail of Sequential GEMOX/NS Chemotherapy in Patients With untreated Pancreatic cancer.

This study aims to evaluate the safety and efficacy of Sequential GEMOX/NS Chemotherapy as a first-line treatment of untreated Pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in the trial and sign the informed consent form
2. 18 years old <age <75 years old
3. Histopathological or cytologically confirmed (inoperable) locally advanced or recurrent metastatic pancreatic ductal adenocarcinoma with lesions measurable according to RECIST criteria
4. ECOG score 0-1
5. Life expectancy > 3 months
6. There must be a CT or MRI examination within a week
7. at least one lesion that can be measured by the RECIST v1.1 standard
8. No chemotherapy has been performed (the interval between postoperative adjuvant chemotherapy must be more than 6 months)
9. without radiation therapy (unless there is at least one measurable target lesion in the non-irradiated area)

Exclusion Criteria:

1. pregnant or lactating women; or those who have fertility but refuse to take contraceptive measures;
2. Severe active infections requiring intravenous antibiotic treatment during enrollment;
3. those who are allergic to the test drug;
4. There is ≥2 neuropathy (CTCAE 4.0);
5. uncontrolled, symptomatic brain metastases or those with a history of uncontrollable psychiatric disorders; severe intellectual or cognitive dysfunction;
6. Congestive heart failure, uncontrollable arrhythmia, myocardial infarction within 6 months, unstable angina, stroke or transient ischemic attack;
7. Have other malignant tumors within 5 years, except for fully treated cervical carcinoma in situ or squamous cell carcinoma of the skin, or basal cell carcinoma of the skin that has been basically controlled;
8. Patients who are unable to follow the protocol or who are unable to follow up;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-01-30 (Estimated); Primary Completion 2020-01-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
PFS | from the first drug administration up to 6 months
  progression-free survival
OS | from the first drug administration up to 1 year
  overall survival